CLINICAL TRIAL: NCT00308919
Title: Phase II Study of Photodynamic Therapy With WST-09 in Patients With Recurrent or Persistent Localized Carcinoma of the Prostate Following Radiation Therapy Failure : Effect of the Light Dose and the Number of Fibres
Brief Title: Study of Photodynamic Therapy in Patients With Prostate Cancer Following Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: STEBA France (Industry)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Steba France
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEC/WST03 658 N/WST 2.08
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-05

CONDITIONS: Recurrent or Persistent Localized Carcinoma of the Prostate Following Radiation Therapy Failure
MeSH Terms: conditions — Recurrence

ARMS (1):
- WST 09 (Experimental): Treatment with WST09 Vascular Photodynamic therapy
  Interventions: Drug: WST09

INTERVENTIONS:
Drug: WST09 — Treatment with WST09 Vascular Photodynamic therapy

SUMMARY:
To assess by MR Imaging the lesions induced by WST09-mediated photodynamic therapy (PDT) in patients with recurrent or persistent localized prostate cancer following definitive radiotherapy using different light doses and multiple illuminating fibres.

DETAILED DESCRIPTION:
Prostate cancer is a leading cause of morbidity and mortality in men around the world. Because of the worldwide increase in life expectancy, a dramatic increase in the number of patients with prostate cancer is expected. It has been estimated that by the year 2002, 92,000 men over 65 years of age were diagnosed annually in the European community, where prostate cancer will account for 12% of all new male cancer diagnoses.

Consequently, radiation therapy is used extensively for primary therapy of prostatic carcinoma. The Management Report of clinically localized prostate cancer by the National Cancer Institute SEER program indicated that 30% of patients choose radiation therapy as their first treatment option. However, the ability of radiation therapy to totally and permanently eradicate prostatic cancer has come under question recently as a result of the high number of patients who have post radiotherapy elevated prostatic specific antigen (PSA) determinations (85%), and the high positive post irradiation biopsy rate (31 90%). With high local recurrence rates possibly influencing death rates, the recurrence of prostate cancer after potentially curative local therapy is becoming a significant urological problem. As patients are being treated for prostate cancer at a younger age, a significant number of them will ultimately fail the primary treatment and will be candidates for safe and potentially curative salvage therapy.

High complication and morbidity rates associated with current salvage therapies demand new and improved means for eradicating recurrent local disease. Photodynamic therapy, which allows the destruction of a tumor by the IV administration of a photosensitizer and the local application of light, may provide such means. Transperineal interstitial photodynamic therapy is a minimally invasive procedure to treat selected patients with failed radiation therapy of prostate cancer. A preliminary phase 1 study using the photosensitizer meso-tetrahydroxyphenyl chlorine (mTHPC) in 14 patients indicated that PDT could produce necrosis in prostate involving cancers recurring after radiotherapy, with a low incidence of complications.

ELIGIBILITY:
- Inclusion Criteria: 18 years of age or older

Ability to understand the patient's information sheet and to give written informed consent

Histologic proof of adenocarcinoma of the prostate 12 months or longer following definitive radiotherapy

Disease confined to the prostate (stage T1-N0 or X-M0 or X or T2-N0 or X -M0 or X) without evidence of regional and/or distant disease

Recent (within 90 days) CT scan of the abdomen and pelvis and radionucleotide bone scan or equivalent radiographic imaging confirming that no disease is outside of the prostate

Recent (within 3 months) cystoscopy if clinically warranted

Serum prostatic specific antigen (PSA) equal to or less than 20 ng/mL

Serum PSA showing two consecutive increases at least 2 weeks apart

Life expectancy more than 5 years, based on co-morbidity not related to prostate cancer

Ability to comply with the requirements of the study

- Exclusion Criteria: Patients who are currently receiving any hormone treatment for prostatic carcinoma or for any other cancer, or have done so within the last 6 months.

Patients who have received or are receiving chemotherapy for prostatic carcinoma or for any other cancer

Patients who are currently receiving any photosensitizing medications (e.g. tetracyclines, sulfonamides, phenothiazines, sulfonylurea hypoglycemic agents, thiazide diuretics and griseofulvin)

Patients who have received a TURP (trans-urethral resection of the prostate)

Patients whose radiation therapy caused extensive cystitis and/or proctitis

Any condition, or history of illness or surgery that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the patient (e.g. significant cardiovascular conditions)

History of non compliance with medical therapy and medical recommendations or an unwillingness or inability to complete patient self-administered questionnaires

Participation in a clinical study or receipt of an investigational treatment within the past 90 days

A history of porphyria

A history of significant allergies, particularly to Cremophor® and Benadryl®

A history of sun hypersensitivity or photosensitive dermatitis

Renal disorders (blood creatinine > 1.5 x ULN)

Hepatic disorders (transaminases > ULN, bilirubin> ULN)

Hematological disorders: (White cells < 2500/mm3, neutrophil< 1500/mm3, platelets <140,000/mm3, Hb < 8 g/dl)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-04; Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Trachtenberg, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Haider MA, Davidson SR, Kale AV, Weersink RA, Evans AJ, Toi A, Gertner MR, Bogaards A, Wilson BC, Chin JL, Elhilali M, Trachtenberg J. Prostate gland: MR imaging appearance after vascular targeted photodynamic therapy with palladium-bacteriopheophorbide. Radiology. 2007 Jul;244(1):196-204. doi: 10.1148/radiol.2441060398. Epub 2007 May 16. PMID 17507719